CLINICAL TRIAL: NCT05322642
Title: Efficacy of the Unified Protocol for Transdiagnostic Treatment for Adolescents With Symptoms of Anxiety and Depression: a School-based Randomized Controlled Trial
Brief Title: Efficacy of the Unified Protocol for the Transdiagnostic Treatment (UP-A; Ehrenreich-May et al., 2018) for Adolescents With Moderate Emotional Symptoms in Educational Settings
Acronym: PSICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eduardo Fonseca Pedrero (Other)
Collaborators: Psicofundación: Fundación Española para Promoción, Desarrollo Científico y Profesional de la Psicolo (Other); Consejo General de la Psicología de España (Unknown)
Responsible Party: Sponsor-Investigator, Eduardo Fonseca Pedrero, Director, University of La Rioja
Organization: University of La Rioja (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Universidad de La Rioja
Record Dates: First submitted 2022-03-15; First posted 2022-04-12 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Anxiety Disorder; Depressive Disorder; Emotional Problem; Emotional Disorder
Keywords: adolescents; depression; anxiety; emotional problems; transdiagnostic; school; evidence-based
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: (UP-A) (Experimental): The UP-A (Ehrenreich et al., 2008) is an emotion-focused, transdiagnostic CBT for adolescents A 10-session youth-focused programmed by adapting the core modules of UP-A, for indicated prevention and school settings.
  Interventions: Behavioral: UPA
- Active control condition (Active Comparator): The active control condition will be based on the 10 session of Progressive Relaxation Training programme of Bernstein and Borkovec.
  It follows a similar structure as the UP-A. A group format will be used.
  Interventions: Behavioral: Active control condition (Progressive Relaxation Training)

INTERVENTIONS:
Behavioral: UPA — UP-A is divided into five main treatment modules and three optional modules. The UP-A seek to positively affect how adolescents with anxiety and/ or depression experiences, think about, and respond to a broad range of negative and positive emotions, rather than disorder-specific emotions (e.g., fear, sadness).
  Arms: Experimental: (UP-A)
Behavioral: Active control condition (Progressive Relaxation Training) — Progressive Relaxation Training (Bernstein and Borkovec) program is divided in ten sessions. Relaxation training often is used in behavior therapy as a means to reduce anxiety, tension, and stress. The goal is to release tension from your muscles, while helping you recognize what that tension feels like.
  Arms: Active control condition

SUMMARY:
The main goal is to assess the efficacy of the Unified Protocol for the Transdiagnostic Treatment (UP-A; Ehrenreich-May et al., 2018) for Adolescents with moderate emotional symptoms in educational settings The goal is to prevent emotional symptoms and improve the socio-emotional adjustment.

DETAILED DESCRIPTION:
Emotional problems, such as anxiety and depression, are among the leading causes of associated disability and burden of disease worldwide among young people. Therefore, it is necessary to address this emerging social challenge through the implementation of prevention strategies in relevant stages of development such as adolescence. In recent years, a transdiagnosis approach to emotional disorders has been promoted, highlighting the unified protocol for transdiagnostic treatment of emotional disorders and symptoms in its different versions (adulthood, adolescence, and childhood). In this context, the main goal is to assess the efficacy of the Unified Protocol for the Transdiagnostic Treatment (UP-A; Ehrenreich-May et al., 2018) for Adolescents with moderate emotional symptoms in educational settings The goal is to prevent emotional symptoms and improve the socio-emotional adjustment. Adolescents aged 12-18 at high risk of for anxiety and depression disorders (cut-off scores 10-15 points, PHQ-9 and GAD-7) are selected. The design is a randomized controlled trial with two groups: active control (relaxation) and experimental (UP-A). Pre-test, post-test, and follow-up at 6, 12 and 18 months will be carried out. The impact of different behavioural, cognitive, affective, social, and academic functioning indicators is analyzed, as well as their effects in the short, medium, and long term. The satisfaction of the program by users (students, parents, and professionals) will also be evaluated. The implementation and validation of manualized and empirically validated psychological intervention programs, such as UP-A, should be a priority in educational and socio-health policies.

ELIGIBILITY:
Inclusion Criteria:

* Be 12-18 years old
* Written informed consent from adolescent and legal guardian
* Being able to understand and read Spanish.
* Moderate depressive and anxiety symptoms according to the screening (score moderate level in the PHQ-9 and GAD-7).

Exclusion Criteria:

* Being diagnosed a mental disorder or alcohol and/or substance dependence disorder.
* The presence of high suicidal risk
* A medical disease or condition which prevent the participant from carry out the psychological treatment.
* Receiving another psychological treatment while the study is still ongoing.
* The increase and/or changes in the medication of participants receiving pharmacological treatment during the study

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms | Baseline to 18 months after start of interventions
  Change in the Patient Health Questionnaire-9 (PHQ-9) total score. PHQ-9 total score for the nine items ranges from 0 to 27.Higher scores mean a worse outcome.
Anxiety symptoms | Baseline to 18 months after start of interventions
  Change in the Generalised Anxiety Disorder Assessment (GAD-7) total score. GAD-7 total score for the seven items ranges from 0 to 21.Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Emotional and behavioural problems | Baseline to 18 months after start of interventions
  Change in the Strengths and Difficulties Questionnaire (SDQ) total score. Total dificulties score range from 0 to 40. Higher scores mean a worse outcome.
Health-related quality of life | Baseline to 18 months after start of interventions
  Change in the Kidscreeen-10 (Health-related quality of life) total score. Total score range from 10 to 50. Higher scores mean a better outcome.
Positive and Negative Affect | Baseline to 18 months after start of interventions
  Change in the Positive and Negative Affect Schedule-Brief child (PANAS-Child brief version) scores. Total scores range (both positive and negative Affect) from 5 to 25. For Positive Affect dimension Higher scores mean a better outcome. For Negative Affect dimension higher scores mean a worse outcome.
Transdiagnostic dimensions | Baseline to 18 months after start of interventions
  Change in Multidimensional Emotional Disorders Inventory (MEDI) scores. Total score range from 0 to 392 Higher scores mean a worse outcome.
Educational achievement outcome | Baseline to 18 months after start of interventions
  Educational outcome measured by grades obtained by participant at school. Range from D to A. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Fonseca Pedrero, PhD, Principal Investigator — University of La Rioja
Locations (1):
- Universidad de la Rioja, Logroño, La Rioja, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Essau CA, Sasagawa S, Jones G, Fernandes B, Ollendick TH. Evaluating the real-world effectiveness of a cognitive behavior therapy-based transdiagnostic program for emotional problems in children in a regular school setting. J Affect Disord. 2019 Jun 15;253:357-365. doi: 10.1016/j.jad.2019.04.036. Epub 2019 Apr 16. PMID 31078836
- [Background] de la Torre-Luque A, Fiol-Veny A, Essau CA, Balle M, Bornas X. Effects of a transdiagnostic cognitive behaviour therapy-based programme on the natural course of anxiety symptoms in adolescence. J Affect Disord. 2020 Mar 1;264:474-482. doi: 10.1016/j.jad.2019.11.078. Epub 2019 Nov 14. PMID 32056776
- [Background] Sandin B, Garcia-Escalera J, Valiente RM, Espinosa V, Chorot P. Clinical Utility of an Internet-Delivered Version of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Adolescents (iUP-A): A Pilot Open Trial. Int J Environ Res Public Health. 2020 Nov 10;17(22):8306. doi: 10.3390/ijerph17228306. PMID 33182711
- [Background] Barlow DH, Harris BA, Eustis EH, Farchione TJ. The unified protocol for transdiagnostic treatment of emotional disorders. World Psychiatry. 2020 Jun;19(2):245-246. doi: 10.1002/wps.20748. No abstract available. PMID 32394551
- [Background] Barlow DH, Farchione TJ, Bullis JR, Gallagher MW, Murray-Latin H, Sauer-Zavala S, Bentley KH, Thompson-Hollands J, Conklin LR, Boswell JF, Ametaj A, Carl JR, Boettcher HT, Cassiello-Robbins C. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders Compared With Diagnosis-Specific Protocols for Anxiety Disorders: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Sep 1;74(9):875-884. doi: 10.1001/jamapsychiatry.2017.2164. PMID 28768327
- [Background] Ehrenreich-May J., Kennedy S.M., Sherman J.A., Bilek E.L., Buzzella B.A., Bennett S.M., Barlow D.H. Unified Protocols for Transdiagnostic Treatment of Emotional Disorders in Children and AdolescentsTherapist Guide: Therapist Guide. Oxford University Press; New York, NY, USA: 2017.